CLINICAL TRIAL: NCT03421912
Title: Comparative Monocentric Randomized Study Evaluating the Satisfaction and Quality of Life of Patients Using Cicaplast Baume B5 Versus Dexeryl for the Management of Cutaneous Toxicities Induced by Epidermal Growth Factor Receptor Inhibitors (iEGRF) in Carcinomas Squamous Cells of the Head and Neck, Colorectal Cancers or Lung Cancers
Brief Title: Satisfaction and Quality of Life Comparison Between Patients Using Cicaplast Baume B5 Versus Dexeryl for the Management of Cutaneous Toxicities Induced by Epidermal Growth Factor Receptor Inhibitors (iEGFR)
Acronym: CICAFIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CICAFIX - ET17-011
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Colorectal Cancer; Non Small Cell Lung Cancer; Epidermal Growth Factor Receptor Inhibitor
Keywords: Prevention strategy; Cutaneous toxicity; Quality of life; Patient satisfaction; Dermatology Life Quality Index (DLQI); Epidermal Repair Score (SCOREPI); Topical treatment
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Arm A : Use of Cicaplast balm B5 since de first day of iEGFR initiation treatment for 30 days Arm B : Use of Dexeryl cream since de first day of iEGFR initiation treatment for 30 days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : Cicaplast balm B5 (Experimental): Use of Cicaplast balm B5, 2 to 3 applications per day, since the first day of iEGFR treatment initiation for 30 days to avoid or limit appearance of cutaneous toxicities related to iEGFR treatment.
  Interventions: Other: Cicaplast Balm B5
- Arm B : Dexeryl (Active Comparator): Use of Dexeryl, 2 to 3 applications per day, since de first day of iEGFR treatment initiation for 30 days to avoid or limit appearence of cutaneous toxicities related to iEGFR treatment.
  Interventions: Other: Dexeryl

INTERVENTIONS:
Other: Cicaplast Balm B5 — The patients have to do 2 to 3 applications per day on the face, on lesions and in poultice in the evening in case of painful crack on the fingers
  Arms: Arm A : Cicaplast balm B5
Other: Dexeryl — The patients have to do 2 to 3 applications per day on the face, on lesions and in poultice in the evening in case of painful crack on the fingers
  Arms: Arm B : Dexeryl

SUMMARY:
This randomized comparative study aims to evaluate the satisfaction and quality of life of patients using Cicaplast balm B5, versus Dexeryl, for the management of cutaneous toxicities of iEGFR in squamous cell carcinoma of the head and neck, cancers colorectal or pulmonary

DETAILED DESCRIPTION:
The arrival of new therapeutic strategies such as targeted therapies has led to real progress in the treatment of cancers. Tyrosine kinase inhibitors and antibodies to epidermal growth factor receptors (EGFR), or iEGFR, target one of the major pathways of tumor cell proliferation. These treatments have demonstrated their interest in the treatment of certain advanced solid malignant tumors (head and neck cancer, colorectal cancer, bronchial cancer).

Although having a much better tolerance profile than the "classical" cytotoxic treatments used in the same indications, these treatments, however, have frequent cutaneous toxicities that are inconvenient for patients. According to the molecules, they can affect 80 to 90% of patients treated from the first weeks of treatment and to different degrees. They appear as well in the skin (acneiform rash, erythema, desquamation, xerosis, pruritus) as skin appendages (paronychia, alopecia).

The consequences of these adverse effects are significant, which may be at the origin of a decrease in dose or even of a stop of anti-tumoral treatment inducing a reduction of the expected clinical benefit. In addition, they represent for the patient a real source of inconvenience and pain, which can impact the quality of life (choice of dress, feeling of shame because of the appearance of the skin ...) and impact the adherence to iEGFR treatment.

Management includes first and foremost preventive measures: the use of moisturizing topicals and dermatological soap-free surgras is recommended as soon as iEGFR treatment is initiated, and preventive systemic treatment with cyclins (doxycycline 100 mg daily) is proposed for at least 6 weeks and then reevaluated for skin toxicity.

In case of appearance of skin toxicities, it is initially prescribed in common practice a topical such as Dexeryl (used in many hospitals as standard) or Cicaplast Balm B5 La Roche Posay (used in current practice at Léon Bérard Center). In a second step, topical corticosteroids are prescribed, depending on the grade of toxicity.

There is, however, no validated argument in the literature to guide the choice of clinicians to use either of these topics. Cicaplast balm B5 (antibacterial, repairing damaged skin, moisturizing and relieving feelings of discomfort) would limit the aggravation of skin toxicities and therefore the use of pharmacological measures, including topical corticosteroids class 3 or 4 may long term, weaken the skin barrier even more.

This randomized comparative study aims to evaluate the satisfaction and quality of life of patients using Cicaplast balm B5, versus Dexeryl, for the management of cutaneous toxicities of iEGFR in squamous cell carcinoma of the head and neck, cancers colorectal or pulmonary

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patient with recurrent and / or metastatic head and neck squamous cell carcinoma OR metastatic colorectal cancer with non-mutated RAS gene (wild-type) OR non-small cell lung cancer (NSCLC) with EGFR activating mutations.
* Treated for the first time by an iEGFR having received a marketing authorization.
* Having signed a consent to participate in the study.
* Affiliated to a health insurance plan (or beneficiary of such a plan).

Exclusion Criteria:

* Concomitant radiotherapy.
* Unresolved skin toxicity from previous treatment, whatever it may be.
* Concomitant use of other topical treatments.
* Known hypersensitivity to at least one of the components of the topicals used.
* Pregnant or lactating women.
* Participation in another clinical trial (even if supportive care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-04-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Overall patient satisfaction after 30 days treatment | After 30 days of treatment or at the end of treatment for patient who interrupt the treatment before 30 days
  Overall patient satisfaction toward Cicaplast balm B5 or Dexeryl will be evaluated by a numerical scale from 0 to 10 in each arm

SECONDARY OUTCOMES:
Overall patient satisfaction after 60 days treatment | After 60 days of treatment or at the end of treatment for patient who interrupt the treatment before 60 days
  Overall patient satisfaction toward Cicaplast balm B5 or Dexeryl will be evaluated by a numerical scale from 0 to 10 in each arm
Patient Quality of life | At inclusion, after 30 and 60 days of treatment
  Quality of life of patient will be evaluated by using the Dermatology Life Quality Index questionnaire (DLQI) in each arm
Cutaneous toxicities evaluation using Epidermal Repair Score (SCOREPI) | After 15, 30 and 60 days of treatment
  Cutaneous toxicities will be evaluated in each arm by using Epidermal Repair Score (SCOREPI)
Cutaneous toxicities evaluation using Common Terminology Criteria for Adverse Events (CTCAE) version 4 | After 15, 30 and 60 days of treatment
  Cutaneous toxicities will be evaluated in each arm by using Common Terminology Criteria for Adverse Events (CTCAE) version 4
Modification/Interruption/Discontinuing iEGFR treatment rate | Continuously up to 30 days after starting treatment
  Modification/Interruption/Discontinuing iEGFR treatment rate in each arm because of cutaneous toxicity
DLQI and SCOREPI scores correlation | After 30 and 60 days of treatment
  Evaluation of DLQI (patient evaluation) and SCOREPI (investigator evaluation) scores correlation in each arm
Topical observance | Between the 1st day and the 15th day of treatment, and between the 15th and the 30th day of treatment
  Topical observance will be evaluated in each arm by data collection by each patient in a diary
Use rate of dermocorticoids | Continously up to 60 days after starting treatment
  Evaluation of the rate of patients needing to use dermocorticoids.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme FAYETTE, Doctor, Principal Investigator — Centre Léon Bérard, Lyon, France
Locations (1):
- Centre Léon Bérard, Lyon, Rhône, France